CLINICAL TRIAL: NCT05960097
Title: A Phase 2 Randomized, Active-controlled, Observer-blind Study to Assess the Safety, Reactogenicity, and Immunogenicity of a Booster Dose of Investigational COVID-19 mRNA Vaccines in Healthy Adults Who Previously Received a Complete Primary Vaccination Series With or Without Booster Dose(s)
Brief Title: A Study on the Safety and Immune Response of Investigational COVID-19 mRNA Vaccines in Healthy Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: CureVac (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 219075
Record Dates: First submitted 2023-07-24; First posted 2023-07-25 (Actual); Results first posted 2025-10-23 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: SARS-CoV-2; COVID-19
Keywords: COVID-19; Pandemic; Booster vaccine
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This is an observer-blind study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Part A: CV0701 mRNA COVID-19 Vaccine (Low dose) (Experimental): Participants received one dose of the CV0701 mRNA COVID-19 vaccine in the low-dose formulation on Day 1.
  Interventions: Biological: CV0701 mRNA COVID-19 Vaccine (Low dose)
- Part A: CV0701 mRNA COVID-19 Vaccine (Medium dose) (Experimental): Participants received one dose of the CV0701 mRNA COVID-19 vaccine in the medium-dose formulation on Day 1.
  Interventions: Biological: CV0701 mRNA COVID-19 Vaccine (Medium dose)
- Part A: CV0701 mRNA COVID-19 Vaccine (High dose) (Experimental): Participants received one dose of the CV0701 mRNA COVID-19 vaccine in the high-dose formulation on Day 1.
  Interventions: Biological: CV0701 mRNA COVID-19 Vaccine (High dose)
- Part A: CV0601 mRNA COVID-19 vaccine (Experimental): Participants received one dose of the CV0601 mRNA COVID-19 vaccine on Day 1.
  Interventions: Biological: CV0601 mRNA COVID-19 Vaccine
- Part A: Control Vaccine (Active Comparator): Participants received one dose of the control vaccine at Day 1.
  Interventions: Biological: Control vaccine
- Part B: CV0801 mRNA COVID-19 vaccine (Maximum storage condition) (Experimental): Participants received one dose of the CV0801 mRNA COVID-19 vaccine on Day 1 under Maximum storage condition.
  Interventions: Biological: CV0801 mRNA COVID-19 Vaccine
- Part B: CV0801 mRNA COVID-19 vaccine (Intermediate storage condition) (Experimental): Participants received one dose of the CV0801 mRNA COVID-19 vaccine on Day 1 under Intermediate storage condition.
  Interventions: Biological: CV0801 mRNA COVID-19 Vaccine
- Part B: CV0801 mRNA COVID-19 vaccine (Baseline-control storage condition) (Experimental): Participants received one dose of the CV0801 mRNA COVID-19 vaccine on Day 1 under Baseline-control storage condition.
  Interventions: Biological: CV0801 mRNA COVID-19 Vaccine

INTERVENTIONS:
Biological: CV0701 mRNA COVID-19 Vaccine (Low dose) — Study vaccine was administered as a single intramuscular injection.
  Arms: Part A: CV0701 mRNA COVID-19 Vaccine (Low dose)
Biological: CV0701 mRNA COVID-19 Vaccine (Medium dose) — Study vaccine was administered as a single intramuscular injection.
  Arms: Part A: CV0701 mRNA COVID-19 Vaccine (Medium dose)
Biological: CV0701 mRNA COVID-19 Vaccine (High dose) — Study vaccine was administered as a single intramuscular injection.
  Arms: Part A: CV0701 mRNA COVID-19 Vaccine (High dose)
Biological: CV0601 mRNA COVID-19 Vaccine — Study vaccine was administered as a single intramuscular injection.
  Arms: Part A: CV0601 mRNA COVID-19 vaccine
Biological: Control vaccine — Study vaccine was administered as a single intramuscular injection.
  Arms: Part A: Control Vaccine
Biological: CV0801 mRNA COVID-19 Vaccine — Study vaccine was administered as a single intramuscular injection.
  Arms: Part B: CV0801 mRNA COVID-19 vaccine (Baseline-control storage condition); Part B: CV0801 mRNA COVID-19 vaccine (Intermediate storage condition); Part B: CV0801 mRNA COVID-19 vaccine (Maximum storage condition)

SUMMARY:
The purpose of Part A of this study is to assess the immune response and safety of a booster dose of investigational COVID-19 mRNA vaccines in healthy adults. The study will compare the investigational vaccines to control vaccine.

The purpose of Part B of this study is to assess the immune response and safety of a booster dose of investigational COVID-19 mRNA vaccines in healthy adults. The study will compare the investigational vaccine under three different storage conditions.

DETAILED DESCRIPTION:
Part A:

This Phase 2 study's Part A evaluates the safety, reactogenicity, and immunogenicity of two candidate vaccines - the bivalent CV0701 and the monovalent CV0601 - in healthy adults who have received a full primary vaccination series (with or without booster doses). By including these candidates, the study will assess whether immune interference occurs between the XY spike protein and the XX spike protein antigens in the bivalent vaccine compared with the XX spike protein antigen in the monovalent vaccine. In Part A, both CV0701 and CV0601 will be compared to the Control Vaccine (that serve as a standard of care control) using a randomized, observer-blinded design.

Part B:

The purpose of Part B is to evaluate the safety and Day 29 immunogenicity of CV0801 under three storage conditions:

* Condition 1: Baseline/control
* Condition 2: Intermediate storage
* Condition 3: Maximum storage

Condition 1 serves as the control against which the performance (safety, reactogenicity, and immunogenicity) of Conditions 2 and 3 will be compared.

mRNA vaccine stability is affected by product-specific factors (e.g., molecular weight, buffer composition, lipid nanoparticle encapsulation), manufacturing factors (such as the duration the vaccine remains in liquid form during production and handling at different temperatures), and storage conditions. The impact of these factors is based on product and process knowledge as well as clinical experience.

Through Part B of this Phase 2 study, GSK and CureVac aim to develop data on how different storage conditions affect the final attributes of the vaccine in a clinical trial setting.

ELIGIBILITY:
Participants are eligible to be included in the study only if all of the following criteria apply:

1. Is at least 18 years old and has achieved legal age according to local regulations in each participating country.
2. Must provide documented informed consent prior to any study procedures being performed.
3. Can and will comply with the requirements of the protocol, in the opinion of the investigator.
4. Is healthy or medically stable as determined by the investigator's judgment based on medical history, vital sign measurements, and physical examination findings. Participants with pre-existing stable disease, defined as disease not requiring significant change in therapy or hospitalization for worsening disease during the 6 weeks before enrollment, can be included.
5. Prior receipt of an mRNA COVID-19 vaccine. This may be from a completed primary vaccination series or booster dose(s) of an approved or authorized mRNA COVID-19 vaccine. The last vaccination must be an mRNA COVID-19 vaccination received at least 3 months prior to randomization.
6. If the participant is a woman of childbearing potential, the participant may be enrolled in the study, if they:

   * have practiced adequate contraception for 30 days prior to study intervention administration; and
   * have a negative pregnancy test result on the day of study intervention administration; and
   * have agreed to continue adequate contraception for 2 months after study intervention administration.

Female participants of non-childbearing potential may be enrolled in the study. Nonchildbearing potential is defined as current salpingectomy, hysterectomy, ovariectomy, or postmenopausal.

Participants are excluded from the study if any of the following criteria apply:

1. Is pregnant or has a positive pregnancy test result at Visit 1.
2. Is breastfeeding or will (re)start breastfeeding from the study intervention administration to 3 months after study intervention administration.
3. Has any medical disease or psychiatric condition that, in the opinion of the investigator, precludes study participation because it would place the participant at an unacceptable risk of injury, would render them unable to meet the requirements of the protocol or may interfere with successful completion of the study.
4. Has any history of an immunosuppressive or immunodeficient condition resulting from disease.
5. Has used immunosuppressants or other immune-modifying drugs for 14 consecutive days or more within 3 months prior to the study intervention administration. Non-systemic corticosteroids are allowed. If systemic corticosteroids have been administered short term (<14 days) for treatment of an acute illness, participants should not be enrolled into the study until corticosteroid therapy has been discontinued for at least 28 days before study intervention administration.
6. Has an acute medical illness or acute febrile illness with oral temperature ≥38.0°C or ≥100.4°F within 72 hours prior to study intervention administration.
7. Has participated in another study involving any investigational product, vaccine, or device within 28 days before the study intervention administration and/or planned participation through end of study (EoS).
8. Has participated in Part A of this study.
9. Has a history of hypersensitivity or severe allergic reaction including anaphylaxis, generalized urticaria, angioedema, and other significant reactions to any previous mRNA vaccine or any component of the study intervention(s).
10. Has received or plans to receive immunoglobulins or any blood or blood products within 3 months before study intervention administration through EoS.
11. Has a bleeding disorder, or prior history of significant bleeding or bruising following intramuscular injections.
12. Has a history of chronic alcohol consumption and/or drug abuse as deemed by the investigator to render the potential participant unable/unlikely to provide accurate safety reports or comply with study procedures.
13. Has a history of myocarditis, pericarditis, or idiopathic cardiomyopathy, or presence of any medical condition that increases risk of myocarditis or pericarditis, including cocaine abuse, cardiomyopathy, endomyocardial fibrosis, hypereosinophilic syndrome, hypersensitivity myocarditis, eosinophilic granulomatosis with polyangiitis and persistent myocardial infection.
14. Has received a live vaccine 30 days before the study intervention administration or has a planned administration within 30 days after the study intervention administration.
15. Has received a non-replicating vaccine 8 days before the study intervention administration or has a planned administration within 14 days after the study intervention administration.
16. Has a documented history of confirmed SARS-CoV-2 infection within 3 months before study intervention administration.
17. Has had known close contact with anyone who had a confirmed SARS-CoV-2 infection within 2 weeks before study intervention administration.
18. Is an employee or family member of the investigator or study site staff.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 692 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (3):
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, Hollywood, Florida
  - GSK Investigational Site, Peoria, Illinois
- Australia (14):
  - GSK Investigational Site, Bruce, Australian Capital Territory
  - GSK Investigational Site, Blacktown, New South Wales
  - GSK Investigational Site, Botany, New South Wales
  - GSK Investigational Site, Brookvale, New South Wales
  - GSK Investigational Site, Coffs Harbour, New South Wales
  - GSK Investigational Site, Darlinghurst, New South Wales
  - GSK Investigational Site, Kanwal, New South Wales
  - GSK Investigational Site, Maroubra, New South Wales
  - GSK Investigational Site, Merewether, New South Wales
  - GSK Investigational Site, Blacktown, Queensland
  - GSK Investigational Site, Sherwood, Queensland
  - GSK Investigational Site, Tarragindi, Queensland
  - GSK Investigational Site, Adelaide, South Australia
  - GSK Investigational Site, Camberwell, Victoria

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: http://www.gsk.com/en-gb/innovation/trials/data-transparency/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 692 participants were included in enrolled set out of which only 686 were included in exposed set and started the study.
Period: Overall Study
Arm/Group | Part A: CV0701 mRNA COVID-19 Vaccine (Low Dose) | Part A: CV0701 mRNA COVID-19 Vaccine (Medium Dose) | Part A: CV0701 mRNA COVID-19 Vaccine (High Dose) | Part A: CV0601 mRNA COVID-19 Vaccine | Part A: Control Vaccine | Part B: CV0801 mRNA COVID-19 Vaccine (Maximum Storage Condition) | Part B: CV0801 mRNA COVID-19 Vaccine (Intermediate Storage Condition) | Part B: CV0801 mRNA COVID-19 Vaccine (Baseline-control Storage Condition)
Started | 87 | 84 | 84 | 85 | 85 | 86 | 87 | 88
Completed | 83 | 83 | 82 | 82 | 83 | 85 | 84 | 85
Not Completed | 4 | 1 | 2 | 3 | 2 | 1 | 3 | 3
Not completed — Lost to Follow-up | 3 | 1 | 1 | 2 | 1 | 1 | 2 | 3
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Early Withdrawal: Participant relocated and cannot attend the site | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: CV0701 mRNA COVID-19 Vaccine (Low Dose) | Part A: CV0701 mRNA COVID-19 Vaccine (Medium Dose) | Part A: CV0701 mRNA COVID-19 Vaccine (High Dose) | Part A: CV0601 mRNA COVID-19 Vaccine | Part A: Control Vaccine | Part B: CV0801 mRNA COVID-19 Vaccine (Maximum Storage Condition) | Part B: CV0801 mRNA COVID-19 Vaccine (Intermediate Storage Condition) | Part B: CV0801 mRNA COVID-19 Vaccine (Baseline-control Storage Condition) | Total
Number analyzed (Participants) | 87 | 84 | 84 | 85 | 85 | 86 | 87 | 88 | 686
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: The Age Continuous analysis is presented separately for Part A and B.
  Years
    Part A: number analyzed (Participants) | 87 | 84 | 84 | 85 | 85 | 0 | 0 | 0 | 425
    Part A | 54.1 (16.71) | 53.3 (16.94) | 52.5 (16.61) | 53.9 (15.53) | 54.2 (16.66) |  |  |  | 53.6 (16.53)
    Part B: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 86 | 87 | 88 | 261
    Part B |  |  |  |  |  | 53.4 (17.94) | 53.2 (17.25) | 54.3 (16.76) | 53.6 (17.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 41 | 37 | 45 | 38 | 42 | 39 | 47 | 334
  Male | 42 | 43 | 47 | 40 | 47 | 44 | 48 | 41 | 352
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Aboriginal Australian | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 4
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Japanese Origin | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 4
  Asian | 6 | 7 | 8 | 7 | 9 | 8 | 11 | 8 | 64
  Black or African American | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 3
  Native Hawaiian or Other Paciﬁc Islander | 1 | 0 | 1 | 3 | 1 | 0 | 1 | 0 | 7
  White | 77 | 76 | 73 | 73 | 73 | 73 | 72 | 76 | 593
  Not Reported | 2 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 6
  Multiple | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 5
  Missing | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Other, Unspecified | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2

OUTCOME MEASURES:

1. Secondary Outcome: Part A: GMT of Serum Neutralization Titers Against Pseudovirus Bearing SARS-CoV-2 Strain XX Spike Protein
Time Frame: At Day 91 and Day 181
Population: Analysis was performed on the PPS which includes all participants from the Exposed Set who were eligible, complied with vaccination as per protocol, and had anti-neutralizing titer against the SARS-CoV-2 strain XX spike protein. Only participants with data available for the specified analysis at the specified timepoints are included.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Part A: CV0701 mRNA COVID-19 Vaccine (Low Dose) | Part A: CV0701 mRNA COVID-19 Vaccine (Medium Dose) | Part A: CV0701 mRNA COVID-19 Vaccine (High Dose) | Part A: CV0601 mRNA COVID-19 Vaccine | Part A: Control Vaccine
Number analyzed (Participants) | 71 | 66 | 73 | 71 | 67
Titers
  Day 91 | 872.5 [686.0 to 1109.7] | 1181.9 [914.8 to 1527.0] | 1477.7 [1160.4 to 1881.8] | 1527.8 [1196.7 to 1950.4] | 1155.6 [896.6 to 1489.3]
  Day 181: number analyzed (Participants) | 59 | 60 | 59 | 59 | 57
  Day 181 | 585.0 [444.3 to 770.3] | 797.0 [600.2 to 1058.5] | 977.6 [738.2 to 1294.6] | 1032.6 [777.1 to 1372.2] | 734.2 [546.9 to 985.7]

2. Secondary Outcome: Part A: GMT of Serum Neutralization Titers Against Pseudovirus Bearing SARS-CoV-2 Strain XY Spike Protein
Time Frame: At Day 91 and Day 181
Population: Analysis was performed on the PPS which includes all participants from the Exposed Set who were eligible, complied with vaccination as per protocol, and had anti-neutralizing titer against the SARS-CoV-2 strain XY spike protein. Only participants with data available for the specified analysis at the specified timepoints are included.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Part A: CV0701 mRNA COVID-19 Vaccine (Low Dose) | Part A: CV0701 mRNA COVID-19 Vaccine (Medium Dose) | Part A: CV0701 mRNA COVID-19 Vaccine (High Dose) | Part A: CV0601 mRNA COVID-19 Vaccine | Part A: Control Vaccine
Number analyzed (Participants) | 71 | 66 | 73 | 71 | 68
Titers
  Day 91 | 2637.0 [2198.6 to 3162.9] | 3714.0 [3058.0 to 4510.8] | 4284.9 [3566.3 to 5148.4] | 3952.1 [3281.3 to 4760.0] | 3216.5 [2656.1 to 3895.1]
  Day 181: number analyzed (Participants) | 59 | 60 | 59 | 59 | 58
  Day 181 | 2215.8 [1779.5 to 2759.0] | 2935.4 [2342.8 to 3677.9] | 3319.3 [2653.8 to 4151.6] | 3243.6 [2584.7 to 4070.5] | 2640.6 [2095.6 to 3327.2]

3. Secondary Outcome: Part A: GMT of Serum Neutralization Titers Against Pseudovirus Bearing SARS-CoV-2 Strain XZ Spike Protein
Time Frame: At Day 29, Day 91 and Day 181
Population: Analysis was performed on the PPS which includes all participants from the Exposed Set who were eligible, complied with vaccination as per protocol, and had anti-neutralizing titer against the SARS-CoV-2 strain XZ spike protein. Only participants with data available for the specified analysis at the specified timepoints are included.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Part A: CV0701 mRNA COVID-19 Vaccine (Low Dose) | Part A: CV0701 mRNA COVID-19 Vaccine (Medium Dose) | Part A: CV0701 mRNA COVID-19 Vaccine (High Dose) | Part A: CV0601 mRNA COVID-19 Vaccine | Part A: Control Vaccine
Number analyzed (Participants) | 78 | 73 | 74 | 74 | 80
Titers
  Day 29 | 196.0 [155.1 to 247.7] | 281.5 [220.6 to 359.3] | 335.0 [262.4 to 427.6] | 404.3 [316.8 to 515.9] | 265.7 [209.2 to 337.5]
  Day 91: number analyzed (Participants) | 71 | 64 | 72 | 71 | 68
  Day 91 | 139.8 [108.1 to 180.9] | 188.6 [142.8 to 249.1] | 259.6 [199.3 to 338.2] | 259.5 [199.6 to 337.2] | 194.5 [148.2 to 255.3]
  Day 181: number analyzed (Participants) | 59 | 59 | 58 | 59 | 58
  Day 181 | 105.3 [78.7 to 140.9] | 131.1 [97.3 to 176.7] | 170.2 [125.7 to 230.5] | 180.2 [133.5 to 243.1] | 117.2 [85.9 to 159.7]

4. Secondary Outcome: Part A: Percentage of Participants With Seroresponse of Serum Neutralization Titers Against Pseudovirus Bearing SARS-CoV-2 Strain XX Spike Protein
Description: Seroresponse is defined as post-booster titer greater than or equal to (≥) 4 times the lower limit of quantification (LLOQ) when pre-vaccination titer is below LLOQ or a post-booster titer ≥ 4 times the pre-booster titer when pre-vaccination titer is ≥ LLOQ.
Time Frame: At Day 29 compared to baseline (Day 1)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part A: CV0701 mRNA COVID-19 Vaccine (Low Dose) | Part A: CV0701 mRNA COVID-19 Vaccine (Medium Dose) | Part A: CV0701 mRNA COVID-19 Vaccine (High Dose) | Part A: CV0601 mRNA COVID-19 Vaccine | Part A: Control Vaccine
Number analyzed (Participants) | 78 | 74 | 75 | 74 | 79
Percentage of participants | 38.5 [27.66 to 50.17] | 50.0 [38.14 to 61.86] | 50.7 [38.86 to 62.42] | 51.4 [39.44 to 63.15] | 48.1 [36.71 to 59.64]

5. Secondary Outcome: Part A: Percentage of Participants With Seroresponse of Serum Neutralization Titers Against Pseudovirus Bearing SARS-CoV-2 Strain XY Spike Protein
Description: Seroresponse is defined as post-booster titer ≥ 4 times the lower limit of quantification (LLOQ) when pre-vaccination titer is below LLOQ or a post-booster titer ≥ 4 times the pre-booster titer when pre-vaccination titer is ≥ LLOQ.
Time Frame: At Day 29 compared to baseline (Day 1)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part A: CV0701 mRNA COVID-19 Vaccine (Low Dose) | Part A: CV0701 mRNA COVID-19 Vaccine (Medium Dose) | Part A: CV0701 mRNA COVID-19 Vaccine (High Dose) | Part A: CV0601 mRNA COVID-19 Vaccine | Part A: Control Vaccine
Number analyzed (Participants) | 78 | 74 | 75 | 74 | 80
Percentage of participants | 17.9 [10.17 to 28.28] | 25.7 [16.22 to 37.16] | 29.3 [19.38 to 40.98] | 25.7 [16.22 to 37.16] | 35.0 [24.67 to 46.48]

6. Secondary Outcome: Part A: Percentage of Participants With Seroresponse of Serum Neutralization Titers Against Pseudovirus Bearing SARS-CoV-2 Strain XZ Spike Protein
Description: Seroresponse is defined as post-booster titer ≥ 4 times the LLOQ when pre-vaccination titer is below LLOQ or a post-booster titer ≥ 4 times the pre-booster titer when pre-vaccination titer is ≥ LLOQ.
Time Frame: At Day 29 compared to baseline (Day 1)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part A: CV0701 mRNA COVID-19 Vaccine (Low Dose) | Part A: CV0701 mRNA COVID-19 Vaccine (Medium Dose) | Part A: CV0701 mRNA COVID-19 Vaccine (High Dose) | Part A: CV0601 mRNA COVID-19 Vaccine | Part A: Control Vaccine
Number analyzed (Participants) | 78 | 73 | 74 | 74 | 80
Percentage of participants | 39.7 [28.83 to 51.46] | 43.8 [32.24 to 55.95] | 55.4 [43.39 to 66.98] | 47.3 [35.57 to 59.25] | 47.5 [36.21 to 58.98]

7. Secondary Outcome: Part A: Geometric Mean Increase (GMI) of Serum Neutralization Titers Against Pseudovirus Bearing SARS-CoV-2 Strain XX Spike Protein
Description: GMI is defined as the the geometric mean of the within participant ratios of the post-dose titer over the pre-dose titer.
Time Frame: At Day 29, Day 91 and Day 181 compared to baseline (Day 1)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Part A: CV0701 mRNA COVID-19 Vaccine (Low Dose) | Part A: CV0701 mRNA COVID-19 Vaccine (Medium Dose) | Part A: CV0701 mRNA COVID-19 Vaccine (High Dose) | Part A: CV0601 mRNA COVID-19 Vaccine | Part A: Control Vaccine
Number analyzed (Participants) | 78 | 74 | 75 | 74 | 79
Ratio
  Day 29 | 2.72 [2.17 to 3.42] | 3.84 [3.03 to 4.87] | 4.56 [3.62 to 5.75] | 4.77 [3.76 to 6.04] | 3.71 [2.94 to 4.68]
  Day 91: number analyzed (Participants) | 71 | 66 | 73 | 71 | 67
  Day 91 | 1.69 [1.33 to 2.15] | 2.29 [1.77 to 2.95] | 2.86 [2.24 to 3.64] | 2.95 [2.31 to 3.77] | 2.23 [1.73 to 2.88]
  Day 181: number analyzed (Participants) | 59 | 60 | 59 | 59 | 57
  Day 181 | 0.96 [0.73 to 1.27] | 1.31 [0.99 to 1.74] | 1.61 [1.21 to 2.13] | 1.70 [1.28 to 2.26] | 1.21 [0.90 to 1.62]

8. Secondary Outcome: Part A: GMI of Serum Neutralization Titers Against Pseudovirus Bearing SARS-CoV-2 Strain XY Spike Protein
Description: as for outcome 7
Time Frame: At Day 29, Day 91 and Day 181 compared to baseline (Day 1)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Part A: CV0701 mRNA COVID-19 Vaccine (Low Dose) | Part A: CV0701 mRNA COVID-19 Vaccine (Medium Dose) | Part A: CV0701 mRNA COVID-19 Vaccine (High Dose) | Part A: CV0601 mRNA COVID-19 Vaccine | Part A: Control Vaccine
Number analyzed (Participants) | 78 | 74 | 75 | 74 | 80
Ratio
  Day 29 | 2.14 [1.79 to 2.55] | 2.68 [2.23 to 3.23] | 3.03 [2.52 to 3.63] | 3.02 [2.51 to 3.63] | 2.79 [2.33 to 3.34]
  Day 91: number analyzed (Participants) | 71 | 66 | 73 | 71 | 68
  Day 91 | 1.41 [1.17 to 1.69] | 1.98 [1.63 to 2.41] | 2.28 [1.90 to 2.75] | 2.11 [1.75 to 2.54] | 1.72 [1.42 to 2.08]
  Day 181: number analyzed (Participants) | 59 | 60 | 59 | 59 | 58
  Day 181 | 1.07 [0.86 to 1.34] | 1.42 [1.14 to 1.78] | 1.61 [1.29 to 2.01] | 1.57 [1.25 to 1.97] | 1.28 [1.02 to 1.61]

9. Secondary Outcome: Part A: GMI of Serum Neutralization Titers Against Pseudovirus Bearing SARS-CoV-2 Strain XZ Spike Protein
Description: as for outcome 7
Time Frame: At Day 29, Day 91 and Day 181 compared to baseline (Day 1)
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Part A: CV0701 mRNA COVID-19 Vaccine (Low Dose) | Part A: CV0701 mRNA COVID-19 Vaccine (Medium Dose) | Part A: CV0701 mRNA COVID-19 Vaccine (High Dose) | Part A: CV0601 mRNA COVID-19 Vaccine | Part A: Control Vaccine
Number analyzed (Participants) | 78 | 73 | 74 | 74 | 80
Ratio
  Day 29 | 2.66 [2.11 to 3.36] | 3.82 [3.00 to 4.88] | 4.55 [3.56 to 5.81] | 5.49 [4.30 to 7.00] | 3.61 [2.84 to 4.58]
  Day 91: number analyzed (Participants) | 71 | 64 | 72 | 71 | 68
  Day 91 | 1.78 [1.37 to 2.30] | 2.40 [1.82 to 3.17] | 3.30 [2.53 to 4.30] | 3.30 [2.54 to 4.29] | 2.47 [1.88 to 3.25]
  Day 181: number analyzed (Participants) | 59 | 59 | 58 | 59 | 58
  Day 181 | 1.16 [0.86 to 1.55] | 1.44 [1.07 to 1.94] | 1.87 [1.38 to 2.53] | 1.98 [1.47 to 2.67] | 1.29 [0.94 to 1.76]

10. Primary Outcome: Part A: Geometric Mean Titer (GMT) of Serum Neutralization Titers Against Pseudovirus Bearing SARS-CoV-2 Strain XX Spike Protein
Time Frame: At Day 29
Population: Analysis was performed on the Per Protocol Set (PPS) which includes all participants from the Exposed Set who were eligible, complied with vaccination as per protocol, and had anti-neutralizing titer against the SARS-CoV-2 strain XX spike protein. Only participants with data available for the specified analysis at the specified timepoints are included.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Part A: CV0701 mRNA COVID-19 Vaccine (Low Dose) | Part A: CV0701 mRNA COVID-19 Vaccine (Medium Dose) | Part A: CV0701 mRNA COVID-19 Vaccine (High Dose) | Part A: CV0601 mRNA COVID-19 Vaccine | Part A: Control Vaccine
Number analyzed (Participants) | 78 | 74 | 75 | 74 | 79
Titers | 1266.7 [1008.1 to 1591.7] | 1786.9 [1409.1 to 2265.9] | 2122.1 [1681.9 to 2677.4] | 2218.6 [1751.4 to 2810.5] | 1725.5 [1367.6 to 2177.0]

11. Primary Outcome: Part A: GMT of Serum Neutralization Titers Against Pseudovirus Bearing SARS-CoV-2 Strain XY Spike Protein
Time Frame: At Day 29
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Part A: CV0701 mRNA COVID-19 Vaccine (Low Dose) | Part A: CV0701 mRNA COVID-19 Vaccine (Medium Dose) | Part A: CV0701 mRNA COVID-19 Vaccine (High Dose) | Part A: CV0601 mRNA COVID-19 Vaccine | Part A: Control Vaccine
Number analyzed (Participants) | 78 | 74 | 75 | 74 | 80
Titers | 3725.0 [3116.4 to 4452.5] | 4680.6 [3886.5 to 5637.0] | 5275.7 [4397.6 to 6329.1] | 5261.2 [4368.3 to 6336.5] | 4863.4 [4058.1 to 5828.5]

12. Primary Outcome: Part B: GMT of Serum Neutralization Titers Against Pseudovirus Bearing SARS-CoV-2 Strain XY Spike Protein
Time Frame: At Day 29
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Part B: CV0801 mRNA COVID-19 Vaccine (Baseline-control Storage Condition) | Part B: CV0801 mRNA COVID-19 Vaccine (Intermediate Storage Condition) | Part B: CV0801 mRNA COVID-19 Vaccine (Maximum Storage Condition)
Number analyzed (Participants) | 77 | 78 | 80
Titers | 5658.8 [4762.8 to 6723.4] | 4889.4 [4097.4 to 5834.5] | 4629.7 [3892.7 to 5506.2]

13. Primary Outcome: Part A: Number of Participants Reporting Any Solicited Administration Site Adverse Events (AEs)
Description: Assessed solicited administration site events included injection site redness (erythema), pain, swelling and lymphadenopathy (defined as localized axillary, cervical or supraclavicular swelling or tenderness ipsilateral to the injection arm). Any = occurrence of the event regardless of intensity grade.
Time Frame: Day 1 to Day 7
Population: Analysis was performed on the eDiary Set which includes all participants in the safety analysis set for whom eDiary data are available post-vaccination for the specified duration.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: CV0701 mRNA COVID-19 Vaccine (Low Dose) | Part A: CV0701 mRNA COVID-19 Vaccine (Medium Dose) | Part A: CV0701 mRNA COVID-19 Vaccine (High Dose) | Part A: CV0601 mRNA COVID-19 Vaccine | Part A: Control Vaccine
Number analyzed (Participants) | 87 | 84 | 84 | 85 | 85
Participants
  Pain | 34 | 46 | 53 | 40 | 54
  Swelling | 0 | 1 | 3 | 1 | 1
  Redness | 2 | 3 | 2 | 1 | 2
  Lymphadenopathy | 7 | 10 | 15 | 12 | 10

14. Primary Outcome: Part A: Number of Participants Reporting Any Solicited Systemic AEs
Description: Assessed solicited systemic events included fever, chills, headache, myalgia (muscle pain), arthralgia (joint pain), and fatigue (tiredness). Fever is defined as body temperature is higher than or equal to (>=) 38ºC; preferred location for measuring the temperature is oral. Any = occurrence of the event regardless of intensity grade.
Time Frame: Day 1 to Day 7
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: CV0701 mRNA COVID-19 Vaccine (Low Dose) | Part A: CV0701 mRNA COVID-19 Vaccine (Medium Dose) | Part A: CV0701 mRNA COVID-19 Vaccine (High Dose) | Part A: CV0601 mRNA COVID-19 Vaccine | Part A: Control Vaccine
Number analyzed (Participants) | 87 | 84 | 84 | 85 | 85
Participants
  Fever | 0 | 1 | 2 | 2 | 3
  Myalgia | 14 | 20 | 35 | 25 | 28
  Chills | 5 | 9 | 11 | 3 | 9
  Fatigue | 30 | 26 | 40 | 24 | 34
  Headache | 20 | 30 | 37 | 27 | 28
  Arthralgia | 9 | 7 | 13 | 4 | 14

15. Primary Outcome: Part A: Number of Participants Reporting Any Unsolicited AEs
Description: An unsolicited AE is an AE that is either not included in the list of solicited events or can be included in the list of solicited events but with an onset outside the specified period of follow-up for solicited events. Unsolicited AEs include both serious and nonserious AEs. Any = occurrence of the event regardless of intensity grade.
Time Frame: Day 1 to Day 28
Population: Analysis was performed on the Exposed Set (ES) which includes all participants who received the study intervention and had unsolicited AEs data available post-vaccination for the specified duration.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: CV0701 mRNA COVID-19 Vaccine (Low Dose) | Part A: CV0701 mRNA COVID-19 Vaccine (Medium Dose) | Part A: CV0701 mRNA COVID-19 Vaccine (High Dose) | Part A: CV0601 mRNA COVID-19 Vaccine | Part A: Control Vaccine
Number analyzed (Participants) | 87 | 84 | 84 | 85 | 85
Participants | 20 | 22 | 21 | 27 | 23

16. Primary Outcome: Part A: Number of Participants Reporting Any Medically Attended Adverse Events (MAAEs), Serious Adverse Events (SAEs) and AEs of Special Interest (AESIs)
Description: An SAE refers to any untoward medical occurrence that results in death, is life-threatening, requires inpatient hospitalization or extends existing hospitalization, causes persistent or significant disability/incapacity, involves a congenital anomaly/birth defect in a participant's offspring, includes an abnormal pregnancy outcome, or occurs in any other situation per the investigator's judgement.
  An MAAE results in a visit to a medical professional, such as televisits, physician's office visits, urgent care visits, emergency rooms visits, or hospitalizations.
  AESIs are severe or non-severe predefined AEs of scientific and medical concern specific to the product/program. This study noted the following AESIs: potential immune-mediated disease (pIMDs), lab-confirmed moderate to severe COVID-19, myocarditis and pericarditis, anaphylaxis, or severe hypersensitivity within 24 hours post-intervention. "Any" indicates the occurrence of the event regardless of its intensity grade.
Time Frame: Day 1 to Day 181
Population: Analysis was performed on the ES which includes all participants who received the study intervention and had post-vaccination data available for the specified duration.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: CV0701 mRNA COVID-19 Vaccine (Low Dose) | Part A: CV0701 mRNA COVID-19 Vaccine (Medium Dose) | Part A: CV0701 mRNA COVID-19 Vaccine (High Dose) | Part A: CV0601 mRNA COVID-19 Vaccine | Part A: Control Vaccine
Number analyzed (Participants) | 87 | 84 | 84 | 85 | 85
Participants
  MAAEs | 29 | 21 | 25 | 31 | 30
  SAEs | 3 | 0 | 3 | 1 | 3
  AESIs | 7 | 2 | 4 | 1 | 5

17. Primary Outcome: Part B: Number of Participants Reporting Any Solicited Administration Site AEs
Description: as for outcome 13
Time Frame: Day 1 to Day 7
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: CV0801 mRNA COVID-19 Vaccine (Maximum Storage Condition) | Part B: CV0801 mRNA COVID-19 Vaccine (Intermediate Storage Condition) | Part B: CV0801 mRNA COVID-19 Vaccine (Baseline-control Storage Condition)
Number analyzed (Participants) | 86 | 87 | 88
Participants
  Pain | 34 | 42 | 42
  Swelling | 3 | 2 | 1
  Redness | 1 | 0 | 3
  Lymphadenopathy | 6 | 5 | 10

18. Primary Outcome: Part B: Number of Participants Reporting Any Solicited Systemic AEs
Description: Assessed solicited systemic events included fever, chills, headache, myalgia (muscle pain), arthralgia (joint pain), and fatigue (tiredness). Fever is defined as body temperature >= 38ºC; preferred location for measuring the temperature is oral. Any = occurrence of the event regardless of intensity grade.
Time Frame: Day 1 to Day 7
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: CV0801 mRNA COVID-19 Vaccine (Maximum Storage Condition) | Part B: CV0801 mRNA COVID-19 Vaccine (Intermediate Storage Condition) | Part B: CV0801 mRNA COVID-19 Vaccine (Baseline-control Storage Condition)
Number analyzed (Participants) | 86 | 87 | 88
Participants
  Fever | 0 | 0 | 0
  Myalgia | 11 | 21 | 19
  Chills | 1 | 2 | 1
  Fatigue | 28 | 28 | 28
  Headache | 19 | 15 | 28
  Arthralgia | 6 | 9 | 9

19. Primary Outcome: Part B: Number of Participants Reporting Any Unsolicited AEs
Description: as for outcome 15
Time Frame: Day 1 to Day 28
Population: Analysis was performed on the ES which includes all participants who received the study intervention and had unsolicited AEs data available post-vaccination for the specified duration.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: CV0801 mRNA COVID-19 Vaccine (Maximum Storage Condition) | Part B: CV0801 mRNA COVID-19 Vaccine (Intermediate Storage Condition) | Part B: CV0801 mRNA COVID-19 Vaccine (Baseline-control Storage Condition)
Number analyzed (Participants) | 86 | 87 | 88
Participants | 17 | 18 | 18

20. Primary Outcome: Part B: Number of Participants Reporting Any MAAEs, SAEs and AESIs
Time Frame: Day 1 to Day 181
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: CV0801 mRNA COVID-19 Vaccine (Maximum Storage Condition) | Part B: CV0801 mRNA COVID-19 Vaccine (Intermediate Storage Condition) | Part B: CV0801 mRNA COVID-19 Vaccine (Baseline-control Storage Condition)
Number analyzed (Participants) | 86 | 87 | 88
Participants
  MAAEs | 24 | 26 | 23
  SAEs | 2 | 2 | 4
  AESIs | 0 | 2 | 2

ADVERSE EVENTS:
Time Frame: Part A and Part B: Solicited AEs from Day 1 to Day 7; Unsolicited AEs from Day 1 to Day 28; SAEs, MAAEs and AESIs from Day 1 to Day 181
Arm/Group | Part A: CV0701 mRNA COVID-19 Vaccine (Low Dose) | Part A: CV0701 mRNA COVID-19 Vaccine (Medium Dose) | Part A: CV0701 mRNA COVID-19 Vaccine (High Dose) | Part A: CV0601 mRNA COVID-19 Vaccine | Part A: Control Vaccine | Part B: CV0801 mRNA COVID-19 Vaccine (Maximum Storage Condition) | Part B: CV0801 mRNA COVID-19 Vaccine (Intermediate Storage Condition) | Part B: CV0801 mRNA COVID-19 Vaccine (Baseline-control Storage Condition)
All-Cause Mortality (participants affected / at risk) | 0/87 | 0/84 | 0/84 | 0/85 | 0/85 | 0/86 | 0/87 | 0/88
Serious Adverse Events (participants affected / at risk) | 3/87 | 0/84 | 3/84 | 1/85 | 3/85 | 2/86 | 2/87 | 4/88
Other Adverse Events (participants affected / at risk) | 64/87 | 68/84 | 72/84 | 62/85 | 75/85 | 62/86 | 55/87 | 65/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: CV0701 mRNA COVID-19 Vaccine (Low Dose) (N=87) | Part A: CV0701 mRNA COVID-19 Vaccine (Medium Dose) (N=84) | Part A: CV0701 mRNA COVID-19 Vaccine (High Dose) (N=84) | Part A: CV0601 mRNA COVID-19 Vaccine (N=85) | Part A: Control Vaccine (N=85) | Part B: CV0801 mRNA COVID-19 Vaccine (Maximum Storage Condition) (N=86) | Part B: CV0801 mRNA COVID-19 Vaccine (Intermediate Storage Condition) (N=87) | Part B: CV0801 mRNA COVID-19 Vaccine (Baseline-control Storage Condition) (N=88)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic cyst (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Endocarditis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ophthalmic herpes simplex (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mixed anxiety and depressive disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endometrial hyperplasia with cellular atypia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: CV0701 mRNA COVID-19 Vaccine (Low Dose) (N=87) | Part A: CV0701 mRNA COVID-19 Vaccine (Medium Dose) (N=84) | Part A: CV0701 mRNA COVID-19 Vaccine (High Dose) (N=84) | Part A: CV0601 mRNA COVID-19 Vaccine (N=85) | Part A: Control Vaccine (N=85) | Part B: CV0801 mRNA COVID-19 Vaccine (Maximum Storage Condition) (N=86) | Part B: CV0801 mRNA COVID-19 Vaccine (Intermediate Storage Condition) (N=87) | Part B: CV0801 mRNA COVID-19 Vaccine (Baseline-control Storage Condition) (N=88)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 7 (7) | 10 (10) | 15 (15) | 12 (12) | 10 (10) | 6 (6) | 5 (5) | 10 (10)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 5 (5) | 9 (9) | 11 (11) | 3 (3) | 9 (9) | 1 (1) | 2 (2) | 1 (1)
Fatigue (General disorders) | 30 (30) | 27 (27) | 40 (40) | 25 (25) | 34 (34) | 28 (28) | 28 (29) | 28 (28)
Fever (General disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 2 (2) | 3 (3) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 3 (3)
Injection site pain (General disorders) | 34 (34) | 46 (46) | 53 (53) | 40 (40) | 54 (54) | 34 (34) | 42 (42) | 42 (42)
Injection site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site swelling (General disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 3 (3) | 2 (2) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Polyp (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site bruise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site haematoma (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 10 (10) | 5 (5) | 8 (8) | 5 (5) | 12 (12) | 4 (4) | 4 (4) | 5 (5)
Carbuncle (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suspected COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syphilis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 5 (6) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 3 (3)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suture related complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendon injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood magnesium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure systolic increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Smear cervix abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitamin D decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (9) | 7 (7) | 14 (14) | 4 (4) | 14 (14) | 6 (6) | 9 (9) | 9 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 14 (14) | 21 (21) | 35 (35) | 25 (25) | 28 (28) | 11 (11) | 21 (21) | 19 (19)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendon pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Disturbance in attention (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 20 (20) | 30 (30) | 37 (37) | 27 (27) | 29 (29) | 19 (19) | 15 (15) | 28 (29)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Transient aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nightmare (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intermenstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail bed bleeding (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2023-09-26): https://cdn.clinicaltrials.gov/large-docs/97/NCT05960097/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-14): https://cdn.clinicaltrials.gov/large-docs/97/NCT05960097/SAP_001.pdf